CLINICAL TRIAL: NCT07249281
Title: Development of MR Microstructural Imaging Markers for Prostate Cancer Diagnosis and Investigation of the Associated Molecular Mechanisms
Brief Title: MR Microstructural Imaging for Prostate Cancer Diagnosis
Status: Recruiting | Type: Observational
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Collaborators: Zhejiang University (Other); Jiangsu Provincial People's Hospital (Other); The First Affiliated Hospital of Dalian Medical University (Other); Zhejiang Hospital (Other); Henan Cancer Hospital (Other Government); Beijing Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: [2025B] IIT.No. 0321
Record Dates: First submitted 2025-09-01; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-08

CONDITIONS: Prostate Cancer; Diffusion MRI
Keywords: Prostate Cancer; Time-dependent Diffusion MRI (TDDMRI); Diagnostic Accuracy; Multi-center Study
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Magnetic Resonance Imaging; Positron-Emission Tomography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — H&E stained histology (biopsy or whole-slide histology) of the prostate tissue for validation of the MRI microstructural features
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prostate Cancer Suspected Cohort: Men with clinical suspicion of prostate cancer who undergo standardized MRI including time-dependent diffusion MRI (TDDMRI). Histopathological confirmation (biopsy or prostatectomy) will be obtained in a subset of participants who provide consent. Diagnostic accuracy of TDDMRI-derived microstructural markers will be evaluated against pathology when available. Participants without pathology will still contribute imaging data for exploratory analyses.
  Interventions: Diagnostic Test: MRI/ MRS (Magnetic Resonance Imaging /Magnetic Resonance Spectroscopy)

INTERVENTIONS:
Diagnostic Test: MRI/ MRS (Magnetic Resonance Imaging /Magnetic Resonance Spectroscopy) — The investigators will compare the diagnostic power of the proposed time-dependent diffusion MRI technique with conventional multiparameter MRI for prostate diagnosis

SUMMARY:
The goal of this multi-center clinical study is to evaluate whether time-dependent diffusion MRI (TDDMRI) can provide reliable microstructural imaging markers for the diagnosis of prostate cancer. The main questions this study aims to answer are:

* Do TDDMRI-derived microstructural parameters (such as cell size and density) improve diagnostic accuracy for prostate cancer compared with conventional MRI?
* How well do the microstructural parameters correlate with whole-slide pathology findings?
* Can the investigators determine diagnostic models combining multiple features for presurgical diagnosis across multiple centers?

Participants with suspected prostate cancer will undergo 3T MRI including TDDMRI. Microstructural parameters will be quantified and compared with standard multiparametric MRI. All participants will also receive prostate biopsy or prostatectomy, and imaging findings will be validated against histopathology.

This study will:

* Collect TDDMRI and conventional MRI data from six hospitals.
* Derive and validate imaging markers of prostate cancer based on microstructural parameters.
* Compare diagnostic performance across centers and against pathology as the reference standard.

DETAILED DESCRIPTION:
Prostate cancer is one of the most common malignancies among men worldwide, and accurate diagnosis is crucial for treatment planning and outcome prediction. Conventional multiparametric MRI (mpMRI) has become an important tool in prostate cancer (PCa) diagnosis; however, its diagnostic performance remains suboptimal, e.g., for differentiating clinically significant from insignificant disease. Time-dependent diffusion MRI (TDDMRI) is an advanced technique that probes water diffusion over different diffusion times, thereby providing sensitivity to tissue microstructural features such as cell size, cellularity, and transmembrane water exchange. These parameters may serve as novel imaging biomarkers for PCa and could improve diagnostic accuracy beyond what is currently achievable with standard MRI techniques.

This is a multi-center diagnostic cohort study with prospective enrollment of suspected PCa participants, along with pathology data. The study is designed to evaluate the clinical utility of TDDMRI for PCa detection, with a focus on developing and validating MR microstructural imaging markers and establish a robust diagnostic model that is generalizable to most clinical settings.

Study Procedures Participants with clinical suspicion of prostate cancer will undergo standardized MRI examinations that include both conventional mpMRI and TDDMRI sequences. Imaging protocols will be harmonized across participating centers to ensure reproducibility of microstructural parameter estimation. Quantitative markers such as cellularity, cell size, and diffusivity metrics will be derived from TDDMRI data.

Histopathological confirmation through prostate biopsy or prostatectomy will be obtained in a subset of participants who provide informed consent. For these cases, imaging-derived microstructural parameters will be directly compared with histological measures. For participants without available pathology, imaging data will still be retained and analyzed for exploratory purposes and for cross-center reproducibility assessments.

Quality Assurance and Data Management

To guarantee data integrity and cross-site consistency, a centralized data management platform will be implemented. Key measures include:

* Predefined imaging protocols and on-site training to minimize variability across centers.
* Automated and manual data validation checks for completeness, range, and logical consistency.
* Periodic source data verification against original imaging files and pathology reports.
* Maintenance of a data dictionary with standardized definitions for all imaging and clinical variables.
* Regular quality control audits and feedback loops to ensure adherence to protocol.

Statistical and Analytical Plan The primary analysis will assess the diagnostic performance of TDDMRI-derived microstructural parameters, with histopathology as the gold standard. Diagnostic metrics including sensitivity, specificity, and the area under the receiver operating characteristic curve (AUC) will be calculated and directly compared with routine mpMRI metrics and PI-RADS scores.

Secondary analyses will evaluate:

* The correlation between TDDMRI biomarkers and Gleason score or tumor cellularity.
* Cross-center reproducibility and robustness of derived biomarkers.
* Subgroup analyses by tumor location, stage, and patient characteristics.
* Exploratory development of diagnostic thresholds or decision rules based on microstructural parameters.

Sample Size and Missing Data The study is planned as a six-center collaborative effort, with an expected 2000 participants. This target sample size accounts for inter-center variability and allows for ~10-15% attrition or unusable imaging. The final dataset is anticipated to include approximately 40% participants with prostate cancer and 60% without, enabling precise estimation of sensitivity and specificity with narrow confidence intervals.

Missing data will be handled according to predefined rules. Incomplete or degraded imaging datasets will be documented and, where possible, analyzed using available sequences.

Overall Aim The overall aim of this study is to validate TDDMRI as a clinically applicable imaging tool and to establish reproducible microstructural imaging markers that can inform prostate cancer diagnosis across diverse clinical settings. By integrating multi-center imaging data with large-scale histopathological validation, this study seeks to advance precision imaging in prostate cancer and provide evidence for the adoption of TDDMRI in routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Clinical suspicion of prostate cancer (elevated PSA, abnormal digital rectal examination, or other clinical indication).
* Undergoing prostate MRI including TDDMRI as part of diagnostic evaluation. Able and willing to provide written informed consent.

Exclusion Criteria:

* Contraindications to MRI (e.g., pacemaker, ferromagnetic implants, severe claustrophobia).
* Prior treatment for prostate cancer (surgery, radiation, hormonal therapy, chemotherapy).
* Severe comorbid conditions precluding MRI or biopsy.
* Inability to provide informed consent.
* Poor image quality due to motion or technical artifacts (assessed at imaging QC).

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Men with clinical suspicion of prostate cancer will be recruited from six participating hospitals. Clinical suspicion may be based on elevated prostate-specific antigen (PSA) levels, abnormal digital rectal examination, or other clinical findings. All participants will undergo prostate MRI including TDDMRI. Histopathological confirmation through biopsy or prostatectomy will be obtained in a subset of participants who consent to tissue sampling. The study population will therefore include both histopathology-positive and -negative cases, enabling evaluation of diagnostic performance and development of imaging-based diagnostic criteria.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Accuracy of TDDMRI for Clinically Significant Prostate Cancer (csPCa) | Within 3 months after MRI and pathology confirmation.
  Area under the receiver operating characteristic curve (AUC, range 0-1; higher values indicate better diagnostic performance) for TDDMRI-derived microstructural parameters to detect csPCa (reference standard: histopathology; Gleason score ≥7).
Development of Imaging-Based Diagnostic Criteria | Within 3 months (at completion of enrollment and pathology confirmation).
  Establishment of threshold values or decision rules for TDDMRI-derived microstructural parameters (e.g., cellularity, cell size index, diffusivity) to differentiate malignant from benign prostate tissue. Diagnostic cutoffs will be derived by ROC analyses and validated against histopathology.

SECONDARY OUTCOMES:
Cross-Center Reproducibility | After completion of enrollment across all centers (up to 24 months).
  Agreement of TDDMRI-derived parameters across participating centers, assessed by intraclass correlation coefficient (ICC; range 0-1, higher indicates better reproducibility).
Sensitivity and Specificity of TDDMRI | Within 3 months after MRI and pathology confirmation.
  Sensitivity and specificity (0-100%; higher indicates better diagnostic performance) of TDDMRI-derived microstructural parameters in identifying clinically significant prostate cancer.
Comparison with Conventional mpMRI | Within 3 months after MRI and pathology confirmation.
  Difference in diagnostic performance (AUC, sensitivity, specificity) between TDDMRI parameters and conventional mpMRI measures : apparent diffusion coefficient (ADC) and Prostate Imaging-Reporting and Data System, version 2.1 (PI-RADS v2.1; score 1-5, higher indicates a higher likelihood of csPCa).
Correlation with Gleason Score | Within 3 months after MRI scan
  Correlation between TDDMRI microstructural parameters (e.g., cellularity, cell size index) and Gleason score from pathology, using Spearman's ρ (range -1 to 1; larger magnitude indicates stronger monotonic association), with 95% confidence intervals.

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - Beijing Hospital, Beijing, Beijing Municipality
  - Henan Cancer Hospital, Affiliated Cancer Hospital of Zhengzhou University, Zhengzhou, Henan
  - The First Affiliated Hospital of Nanjing Medical University (Jiangsu Province Hospital), Nanjing, Jiangsu
  - The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided
The investigators will share the study protocol after its publication